CLINICAL TRIAL: NCT03098615
Title: An Investigator Initiated Pilot Study Evaluating the Efficacy of Efinaconazole 10% Solution (Jublia) for the Treatment of Onychomycosis With Dermatophytomas
Brief Title: Study Evaluating the Effect of Jublia on Dermatophytomas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Boni Elewski, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F150408010
Record Dates: First submitted 2015-10-16; First posted 2017-04-04 (Actual); Results first posted 2019-03-19 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Onychomycosis; Dermatophytosis
MeSH Terms: conditions — Onychomycosis; Tinea | interventions — efinaconazole; Solutions

STUDY DESIGN:
Intervention Model Description: Topical application of Jublia (Efinaconazole 10% Topical Solution) to patients with distal lateral subungual onychomycosis with dermatophytoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Jublia (Efinaconazole 10% Topical Solution) + nail polish (Other): Subjects with distal lateral subungual onychomycosis (DLSO) with dermatophytoma.
  Interventions: Drug: Jublia (Efinaconazole 10% Topical Solution)

INTERVENTIONS:
Drug: Jublia (Efinaconazole 10% Topical Solution) — Efinaconazole 10% Topical Solution will be applied to the great toenail with the DLSO and dermatophytoma.
  Other Names: Jublia

SUMMARY:
This study will examine how Jublia affects dermatophytomas, which are difficult to treat with other therapeutic options.

DETAILED DESCRIPTION:
Dermatophytomas are known to be resistant to even long courses of systemic antifungals, and have therefore been excluded from both topical and systemic clinical trials for onychomycosis, including those for Efinaconazole solution. Efinaconazole (Jublia) 10% solution is an FDA approved topical medication indicated for treatment of distal lateral subungual onychomycosis (DLSO), and the utility of this medication likely exceeds published results. Efinaconazole solution's novel ability to penetrate into the subungual space likely accounts for improved treatment results seen in DLSO treated with Jublia. We will investigate the utility of topical efinaconazole solution in the treatment of dermatophytomas.

ELIGIBILITY:
Inclusion Criteria:

* Has the informed consent been signed and patient's questions answered.
* Age >= 18
* Patient willing and able to participate for the full duration of the study
* No onychomycosis
* Greater than 4 weeks from prior major surgery for any indication
* Willing to abstain from:

The application of other topical medications or cosmetic products to the toenail Professional pedicures for the duration of the study. - Females of childbearing potential must: Have been using adequate contraception (abstinence, intrauterine device (IUD), birth control pills or spermicidal gel with diaphragm or condom) since their last menses Agree to continue using adequate means of contraception (abstinence, IUD, birth control pills or spermicidal gel with diaphragm or condom) for the duration of study participation

Females are not considered to be of childbearing potential if they are at least 1 year postmenopausal or have had a tubal ligation, bilateral oophorectomy or hysterectomy.

Exclusion Criteria:

* Active onychomycosis of the toenails or fingernails
* Any of the following in the 4 weeks (or as indicated) prior to randomization:

Major surgery for any indication

- Any personal history of: Invasive cancer diagnosed or treated within the past 5 years. Participants who have been in remission for 5 years or more and have not required treatment in the past 5 years may be eligible if the principal investigator believes there is little to no risk of recurrence.

* Concurrent use of the following medications or treatments Other topical antifungals for any concomitant infection
* Females who are pregnant or lactating. Should a woman become pregnant or suspect she is pregnant while she is participating in this study she should notify the study physician immediately.
* Uncontrolled concurrent illness including ongoing or active infection, psychiatric illness/social situations that would limit compliance with study requirements or other underlying serious medical condition which, in the investigator's opinion, might preclude study participation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boni E Elewski, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Jublia Treatment Group: The intervention to be administered is Jublia (Efinaconazole 10% Topical Solution). The frequency of administration is daily to the affected toes.
Period: Overall Study
Arm/Group | Jublia Treatment Group
Started | 19
Completed | 17
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Baseline Group: Subject with age >18, provision of informed consent, presence of dermatophytoma on one or both great toenails, target great to-nail thickness <= 3.0 mm, positive potassium hydroxide (KOH) or culture. Exclusion based upon history of immunosuppression, history of psoriasis of the nail, other nail disease, 3 or more dermatophytomas, unwillingness to avoid nail polish
Arm/Group | Baseline Group
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Elimination of Dermatophytomas That Occur in Distal Lateral Subungual Onychomycosis (DLSO)
Description: Clear nail growth between the proximal nail fold and the dermatophytoma's proximal edge will be measured.
Time Frame: week 48
Measure: Count of Participants; unit: Participants
Groups:
- Baseline Group: Subject with age >18, provision of informed consent, presence of dermatophytoma on one or both great toenails, target great to-nail thickness <= 3.0 mm, positive KOH or culture. Exclusion based upon history of immunosuppression, history of psoriasis of the nail, other nail disease, 3 or more dermatophytomas, unwillingness to avoid nail polish.
Arm/Group | Baseline Group
Number analyzed (Participants) | 19
Participants | 19

2. Secondary Outcome: Clinical or Mycological Cure of Nail
Description: Completely normal nail plate or negative fungal culture
Time Frame: week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Jublia (Efinaconazole 10% Topical Solution) + Nail Polish
Number analyzed (Participants) | 19
Participants | 12

ADVERSE EVENTS:
Time Frame: 48 months
Arm/Group | Baseline Group
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT03098615/Prot_SAP_000.pdf